CLINICAL TRIAL: NCT07155785
Title: The Role of Lidocaine Spray in Reducing Pain During Intrauterine Device Application
Acronym: Lidocaine IUD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Ergul Demircivi Bor, assistant professor, Istanbul Medeniyet University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2022-0285
Record Dates: First submitted 2024-03-13; First posted 2025-09-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Intrauterine Device Migration; Pain
Keywords: intrauterine device; pain
MeSH Terms: conditions — Intrauterine Device Migration; Pain

STUDY DESIGN:
Intervention Model Description: double blind randomized controlled study
Who Masked: Participant, Care Provider, Investigator
Masking Description: off labeled and hidden bottle usage during spray apply
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active group (Active Comparator): This group received lidocaine spray during intrauterine device application.
  Interventions: Drug: Lidocain spray
- Placebo group (Placebo Comparator): This group received saline spray during intrauterine device application.
  Interventions: Drug: Lidocain spray

INTERVENTIONS:
Drug: Lidocain spray — Lidocaine spray as a local anaesthetic agent was applied to the cervix before intrauterine device application.

SUMMARY:
Investigators aimed to investigate the effectiveness of the use of local lidocaine spray application to make routine intrauterine intrauterine device application more painless.

DETAILED DESCRIPTION:
As a standard, no anaesthesia is applied to the patient during intrauterine device application in outpatient clinic conditions. Patients can usually tolerate the procedure even if there is minimal pain and discomfort. In patients with low pain tolerance, the procedure can be terminated before the application can be performed and the application can be repeated under local or general anaesthesia. Local anaesthetic sprays are routinely and comfortably used in episiotomy repair, upper gastrointestinal tract endoscopy and intraoral procedures. In our study, investigators aimed to demonstrate the efficacy of local spray anaesthesia without side effects for the relief of pain that occurs in some patients during intrauterine device application by comparing it with placebo.

ELIGIBILITY:
Inclusion Criteria:

* 18-45 years old patient who comes to have an intrauterine device inserted voluntarily
* The patient who gave consent to participate in the study

Exclusion Criteria:

* Patients who cannot have an intrauterine device because of fibroids or cervical stenosis
* Patient who did not want to participate in the study

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-02-20 (Actual); Study Completion 2023-05-25 (Actual)

PRIMARY OUTCOMES:
Pain component | 1 hour
  Reduction of the pain felt during application of the intrauterine device

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medeniyet University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Only the results of the patients can be shared